CLINICAL TRIAL: NCT00210548
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Dose-Response Study to Evaluate the Efficacy and Safety of 3 Fixed Doses (50 mg eq., 100 mg eq., and 150 mg eq.) of Paliperidone Palmitate in Subjects With Schizophrenia
Brief Title: A Study to Evaluate the Effectiveness and Safety of 3 Doses of Paliperidone Palmitate in Treating Subjects With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR002353; NCT00147173 (obsolete NCT alias)
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2010-04

CONDITIONS: Schizophrenia
Keywords: schizophrenia; intramuscular injection; antipsychotic agents; dementia praecox; paliperidone palmitate; mental disorders; PANSS.
MeSH Terms: conditions — Schizophrenia; Mental Disorders | interventions — Paliperidone Palmitate

INTERVENTIONS:
Drug: paliperidone palmitate

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of 3 doses of paliperidone palmitate in treating subjects with schizophrenia.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, parallel-group, multicenter, dose-response study of patients who have a Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM IV) diagnosis of schizophrenia. The duration of the study is approximately 14 weeks, including a screening period of 1 week and a 13-week double-blind treatment period. Efficacy and safety will be evaluated periodically throughout the study. Samples for pharmacokinetic evaluation will be collected at designated time points, and a blood sample will be collected at baseline (before the start of double-blind treatment) for an optional pharmacogenomics (genetics) analysis. The hypothesis is that the 3 fixed doses of paliperidone are each more efficacious than placebo in treating subjects with schizophrenia. The effectiveness is measured primarily by the change in the Positive and Negative Syndrome Scale for Schizophrenia (PANSS), and secondarily, by the investigator's Clinical Global Impression of Severity (CGI-S) and by the investigator's evaluation of the patient on a Personal and Social Performance (PSP) Scale. Four injections of paliperidone palmitate 50, 100, or 150 milligrams equivalent administered in the gluteal muscle (buttocks). Injections will be given on Days 1, 8, 36, and 64 of the double-blind treatment period of the study.

ELIGIBILITY:
Inclusion Criteria:

* A DSM-IV diagnosis of schizophrenia (disorganized, catatonic, paranoid, residual, or undifferentiated type) for at least 1 year before the screening evaluation
* a total PANSS score of 70 to 120 at screening and baseline (pre-treatment) evaluations
* a body mass index (BMI [weight (kilograms)]/[height (meters)]²) of more than 17.0 kg/m²

Exclusion Criteria:

* A primary active DSM-IV Axis I diagnosis other than schizophrenia
* a decrease of 25% or more in the total PANSS score between screening and baseline evaluations
* a DSM-IV diagnosis of active substance dependence within 3 months of screening evaluation
* a history of treatment resistance as defined by failure to respond to 2 adequate trials of different antipsychotic medications
* a woman who is pregnant, breast-feeding, or planning to become pregnant during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 366 (Actual)
Dates: Start 2005-04; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
The change in the total score of the Positive and Negative Syndrome Scale for Schizophrenia (PANSS) from the beginning to the end of the double-blind treatment period or to the last post-randomization assessment.

SECONDARY OUTCOMES:
The investigator's Clinical Global Impression of the Severity (CGI-S) of schizophrenia and rating of mental function on a Personal and Social Performance Scale (PSP). Evaluations of adverse events, laboratory tests, and other measures of drug safety.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Derived] Gopal S, Hough DW, Xu H, Lull JM, Gassmann-Mayer C, Remmerie BM, Eerdekens MH, Brown DW. Efficacy and safety of paliperidone palmitate in adult patients with acutely symptomatic schizophrenia: a randomized, double-blind, placebo-controlled, dose-response study. Int Clin Psychopharmacol. 2010 Sep;25(5):247-56. doi: 10.1097/YIC.0b013e32833948fa. PMID 20389255
- See also: A study to evaluate the efficacy and safety of 3 doses of paliperidone palmitate in treating subjects with schizophrenia — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=470&filename=CR002353_CSR.pdf